CLINICAL TRIAL: NCT02716519
Title: Clinical Outcomes for Chronic Ulcers Treated With Clostridial Collagenase (SANTYL®) Versus Standard Care Within the Continuum of Care of an Accountable Care Organization (ACO)
Brief Title: Use of Santyl Within an Accountable Care Organization
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017-101-09-037
Record Dates: First submitted 2016-03-02; First posted 2016-03-23 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Pressure Ulcer; Foot Ulcer, Diabetic
Keywords: Diabetes; diabetic foot ulcer; foot sore; type 2 diabetes; type 1 diabetes; DFU; pressure ulcers; bed sores
MeSH Terms: conditions — Pressure Ulcer; Diabetic Foot; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1 | interventions — Collagenases; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Santyl (Experimental): Collagenase ointment applied topically once per day for up to six weeks
  Interventions: Biological: Santyl
- Standard Card (Active Comparator): Standard Care not specified by the protocol; Investigators choose the appropriate standard care treatment for each participant
  Interventions: Other: Standard Care

INTERVENTIONS:
Biological: Santyl — Collagenase ointment applied topically once per day for up to six weeks
  Arms: Santyl
Other: Standard Care — Standard Care not specified by the protocol; Investigators choose the appropriate standard care treatment for each participant
  Arms: Standard Card

SUMMARY:
This study is designed to assess the comparative effectiveness of SANTYL® versus standard of care in the treatment of pressure ulcers and diabetic foot ulcers within the continuum of care of an ACO. After meeting study criteria, participants will be randomly assigned to apply Santyl or standard care to their pressure ulcer or diabetic foot ulcer for up to 6 weeks. Participants will be followed for one year from the date of randomization to assess ulcer status and ulcer complications.

ELIGIBILITY:
INCLUSION CRITERIA

1. Provide written informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information.
2. Eighteen (18) years of age or older, of either sex, and of any race or skin type.
3. Willing and able to make all required study visits.
4. Able to follow instructions and perform the dressing changes at home or have a caregiver who can perform the dressing changes according to the protocol.
5. Subject is currently being treated in an in-patient acute care setting.
6. Willing to use an appropriate off-loading device to keep weight off of foot ulcers; currently receiving adequate pressure redistribution according to local protocol in the affected area for pressure ulcers.
7. For DFU: An ulcer present on any part of the plantar surface of the foot or plantar surface of the hallux which is 0.5 cm2 - 10 cm2 inclusive (as measured at the Screening Visit using the ARANZ Silhouette imaging device).

   For PU: Stage II-IV ulcer that is 1 cm2 to 64 cm2 inclusive (as measured at the Screening Visit using the ARANZ Silhouette imaging device).

   - Subjects may have more than one ulcer without limitation on the ulcer burden, but only one qualifying ulcer per subject will be selected for the study (selection based on greatest clinical need, as determined by the Investigator).
8. For lower extremity ulcers: Adequate arterial blood flow as evidenced by an ankle brachial index (ABI) of > 0.70 and ≤ 1.2. If ABI > 1.2, perfusion at or near the site of the ulcer must be confirmed: i.e., the foot is warm to the touch and has palpable pulses. Availability of an ABI completed within the 90 days of Screening is acceptable.
9. Separation of at least 5 cm (closest ulcer edge to other closest ulcer edge) as measured using the ARANZ Silhouette imaging device if ≥ 2 ulcers are present.
10. Target ulcer is not infected based on clinical assessment.

EXCLUSION CRITERIA

1. Contraindications or hypersensitivity to the use of clostridial collagenase.
2. Participation in another clinical trial within thirty (30) days of Screening, or planned participation overlapping with this study.
3. Bleeding disorder that would preclude sharp debridement during the study.
4. Active cellulitis of the target ulcer, lymphangitic streaking, deep tissue abscess, or infection of muscle, tendon, joint or bone.
5. Co-morbidities leading to systemic organ dysfunction or severe single- or multi-organ failure that in the opinion of the Investigator would preclude safe subject participation in the study.
6. A target ulcer which involves the underlying tissues of tendon.
7. Diagnosis of chronic granulomatous disease, leukocyte adhesion defects, or severe neutropenia.
8. Current treatment (at the time of the Screening Visit) with any of the following:

   * Systemic corticosteroids. If corticosteroid treatment was for ≥ 10 days, there must be a 1 week interval between discontinuation and screening.
   * Immunosuppressive agents
   * Chemotherapeutic agents
   * Antiviral agents
   * Systemic antibiotic therapy for acute wound-related infection
   * Topical antibiotic treatment of the target ulcer
9. Treatment of target ulcer with bioactive therapies within 1 month of screening:

   * Platelet-derived growth factor (e.g., Regranex)
   * Cellular or Tissue-based Products (e.g., Apligraf, Dermagraft, Integra, Oasis, etc.)
   * Amniotic membrane products (e.g., EpiFix, Grafix, etc.)
10. Prior treatment of target ulcer for any length of time with CCO (SANTYL) within 30 days of screening.
11. Any prior radiation therapy to the affected area
12. Medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.
13. Blood counts and blood chemistry values as follows:

NOTE: Availability of lab results within the 30 days of Screening is acceptable.

* Alanine aminotransferase (ALT) > 3x upper limit of normal
* Aspartate aminotransferase (AST) > 3x upper limit of normal
* Gamma Glutamyl Transferase (GGT) > 2.5x upper limit of normal
* Serum albumin < 2.0 g/dL
* Pre-albumin levels of < 10 mg/dL
* Alkaline phosphatase > 500 U/L
* Serum total bilirubin > 3.0 mg/dL
* Serum BUN > 75 mg/dL
* Serum creatinine > 4.5 mg/dL
* HbA1c > 12%
* Hemoglobin (Hgb) < 8.0 g/dL
* WBC < 2.0 x 109/L
* Absolute neutrophil count < 1.0 x 109/L
* Platelet count < 50 x 109/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Target Ulcer Complications | 12 months
  Target ulcer complications from baseline to the end of the assessment period in each treatment group:
  * increase in size by more than 25%,
  * cellulitis,
  * ulcer infections,
  * osteomyelitis,
  * requirement for surgical intervention

SECONDARY OUTCOMES:
The incidence of increase in ulcer size by more than 25% between treatment groups during the assessment period | 12 months
The incidence of cellulitis between treatment groups during the assessment period | 12 months
The incidence of ulcer infections between treatment groups during the assessment period | 12 months
The incidence of osteomyelitis between treatment groups during the assessment period | 12 months
The incidence of requirement for surgical intervention between treatment groups during the assessment period | 12 months
Percentage change in ulcer area from baseline to the end of treatment period | 12 months
Study discontinuations (target ulcer related) | 12 months
Hospital readmission for target ulcer treatment | 12 months
Emergency department visits for target ulcer treatment | 12 months
During the acute phase, daily time at bedside for target ulcer treatment | 6 months
During the acute phase, daily wound care products (including dressings) for target ulcer treatment | 6 months
  During the acute phase, the quantity of daily wound care products (including dressings) for target ulcer treatment will be collected. At the conclusion of the study, the wound care products used will be costed using national costing averages. Total costs will be aggregated on a per patient basis and then compared between the standard of care group and the Santyl group.
During the acute phase, daily antibiotics and analgesics used for target ulcer treatment | 6 months
During the acute phase, daily lab tests for target ulcer treatment | 6 months
During the acute phase, daily surgical procedures for target ulcer treatment | 6 months
During the post-acute phase, weekly clinician time at bedside for target ulcer treatment | 12 months
During the post-acute phase, weekly patient and caregiver time for target ulcer treatment | 6 months
During the post-acute phase, weekly wound care products (including dressings) for target ulcer treatment | 6 months
During the post-acute phase, weekly antibiotics and analgesics used for target ulcer treatment | 6 months
During the post-acute phase, weekly lab tests for target ulcer treatment | 6 months
During the post-acute phase, weekly surgical procedures for target ulcer treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaime E Dickerson, PhD, Study Chair — Smith & Nephew, Inc.; Sandeep Kathju, MD/PhD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes